CLINICAL TRIAL: NCT07031154
Title: A Single-arm, Multicenter, Prospective Clinical Study of Adebrelimab Combined With Apatinib Neoadjuvant Therapy for Resectable Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL-2024KY236-01
Record Dates: First submitted 2025-05-21; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-02

CONDITIONS: Non-Small Cell Lung Cancer; Adebrelimab; Apatinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adebrelimab in combination Apatinib (Experimental)
  Interventions: Drug: Adebrelimab; Drug: Apatinib

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab 1200mg, iv, D1，Q3W
Drug: Apatinib — Apatinib 250mg，P.O，qd，Q3W

SUMMARY:
To evaluate the major pathological response rate of Adibelimab combined with Apatinib neoadjuvant therapy in resectable non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria to be enrolled in the study:
* 18 years old ≤ age ≤70 years old, male or female;
* ECOG PS score 0-1;
* Patients who have not received systematic treatment before and agree to receive radical surgical treatment; Thoracic surgeons judge patients with no contraindications to surgery;
* Stage II, IIIA, or selective stage IIIB (T3N2M0 only) squamous cell or non-squamous non-small cell lung cancer confirmed by histopathology or cytology and determined by the investigator to be capable of R0 resection for curative purposes. Staging should be based on the American Joint Committee on Cancer (AJCC)/Union International Against Cancer (UICC) NSCLC Staging System Version 8;

  1. Not allowed to invade the heart, great blood vessels, trachea, recurrent laryngeal nerve, esophagus, vertebrae, protuberances,And T4 tumors with dispersed tumor nodules in different lung lobes on the same side;
  2. Upper lung groove cancer is not allowed;N2 was defined as mediastinal lymph node non-giant metastases (lymph node diameter < 2cm) confirmed by imaging or pathology and expected to be completely resectable.
* There were enough tumor tissues to detect PD-L1 expression and PD-L1 ≥1%;
* At least one measurable lesion (according to RECIST 1.1 criteria);
* Expected survival of at least 12 weeks;
* Other major organs (liver, kidney, blood system, etc.) function well:

  1. Hemoglobin ≥90g/L (no blood transfusion, no hematopoietic factors, and no drug correction within 2 weeks prior to the first dose);Absolute neutrophil count (ANC) ≥1.5×109/L;
  2. Platelet count ≥100×109/L;
  3. Total bilirubin ≤1.5 times the upper limit of normal value;
  4. Alanine aminotransferase, ASpartate aminotransferase, alkaline phosphatase ≤2.5 times the upper limit of normal value;
  5. Serum creatinine ≤1.5 times the upper limit of normal value; And endogenous creatinine clearance ≥60ml/min;
  6. International Standardized Ratio of prothrombin time (INR)≤1.5 and activated partial thromboplastin time (APTT)≤1.5 times the upper limit of normal for patients who have not received anticoagulant therapy.
* No systemic metastasis (including M1a, M1b, M1c);
* Complete excision is expected;
* Lung function is good and can tolerate surgical treatment;
* Fertile female subjects must have a negative pregnancy test (serum or urine) within 3 days prior to the start of the study drug, and be willing to use a medically approved highly effective contraceptive during the study period and 90 days after the last study drug administration(e.g. intrauterine devices, contraceptives, or condoms); Male subjects whose partner is a woman of reproductive age must consent to use effective contraception or have been surgically sterilized during the study period and 90 days after the last study dosing;
* Subjects voluntarily participate in this clinical study and sign informed consent.

Exclusion Criteria:

* Subjects will not be admitted to the study if they have any of the following conditions:
* have received any anti-tumor therapy in the past, including radiotherapy, chemotherapy, immunotherapy and traditional Chinese medicine anti-tumor therapy (except the treatment of malignant tumors with radical treatment and no recurrence and metastasis for more than 5 years);
* Subjects with non-squamous cell histological types of NSCLC with EGFR mutation positive or ALK positive. Non-squamous cell carcinoma subjects must undergo EGFR gene testing and ALK gene and/or immunohistochemical testing;
* Patients with distant metastases (including M1a, M1b, and M1c);
* Have any active autoimmune disease or history of autoimmune disease (such as uveitis, enteritis, hepatitis, pituitaritis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (may be included after hormone replacement therapy), tuberculosis); Skin conditions (such as vitiligo, psoriasis, or alopecia) with complete remission of childhood asthma that do not require any intervention in adulthood and do not require systemic treatment may be included, but patients requiring medical intervention with bronchodilators may not be included;
* Exclude evidence of past or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiological pneumonia, drug-induced pneumonia, radiographic evidence of active pneumonia, and severe impairment of lung function;
* Subjects who have received systemic treatment with corticosteroids (>10 mg/ day of prednisone or other equivalent hormones) or other immunosuppressants within 2 weeks prior to initial dosing. In the absence of active autoimmune disease, inhaled or topical corticosteroids are permitted, as well as adrenal hormone replacement therapy at doses ≤10 mg/ day of prednisone efficacy;
* Imaging (CT or MRI) shows that the tumor has invaded large blood vessels or the boundary with blood vessels is blurred; Or imaging (CT or MRI) showing the presence of any pulmonary cavities or necrotic lesions, as determined by the investigator;
* Patients who had experienced arteriovenous thrombosis events, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism within 6 months before enrollment;
* Had clinically significant bleeding symptoms or definite bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, etc., or were receiving thrombolytic or anticoagulant therapy within 3 months before enrollment;
* Obvious symptoms of hemoptysis or daily hemoptysis volume of 2.5mL or more within 1 month before enrollment;
* Patients with hypertension who are not well controlled by antihypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg); Or grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥450ms in men and women)≥470ms); According to NYHA criteria, patients with grade Ⅲ to Ⅳ cardiac insufficiency or left ventricular ejection fraction (LVEF) < 50% indicated by cardiac color ultrasound;
* Major operations or serious external injuries of other systems were performed within 2 months before the start of the study;
* Urine routine indicated urinary protein ≥(++), or 24h urinary protein ≥1g or severe hepatic and renal insufficiency;
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
* Allergic to the experimental drug;
* Co-existing with HIV infection or active viral hepatitis;
* Pregnant or lactating women; The fertile subject is unwilling or unable to take effective contraceptive measures;
* Those who suffer from neurological diseases or mental diseases and cannot cooperate;
* Other malignancies developed within 5 or less years before admission, excluding adequately treatable cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery;
* Other situations deemed unsuitable for inclusion by the researcher.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (MPR) | Four weeks after surgery
  When the tumor was surgically resected, the active tumor tissue in the surgical specimen was less than 10%

SECONDARY OUTCOMES:
Pathological complete response (pCR) | Four weeks after surgery
R0 resection rate | Four weeks after surgery
Objective response rate (ORR) | Up to 3 months per 2 cycles (21 days per cycle)
The incidence of adverse events (including serious adverse events) and rank | Up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No